CLINICAL TRIAL: NCT02623400
Title: The Effect of Perinatal Stress on the Development of Preterm Infants
Acronym: RESILIENCE
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S58807
Record Dates: First submitted 2015-11-23; First posted 2015-12-07 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Premature Birth of Newborn
Keywords: preterm birth; perinatal stress; growth and development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva samples of both parents and the child, blood sample of mother and child, cord blood sample,
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infants and their parents: Preterm infants born before 34 weeks gestational age and/or with a birth weight lower than 1500g and their parents.

SUMMARY:
In this project, the investigators will study a cohort of preterm infants, together with their parents, during NICU hospitalization and follow their developmental trajectory until the age of two.

An important first scientific goal of the project is to identify objective stress markers that can be obtained easily and non-invasively in preterm infants during NICU hospitalization. This will include the development of novel techniques to measure stress related heart rate variability (HRV) and EEG maturation, as well as sleep stage markers for preterm infants.

Secondly, the investigators will study the emotional and bonding processes in parents of preterm infants. Parental distress in terms of depressive symptoms, anxiety, perceived stress and parent-infant bonding will be measured at multiple measuring points. This will enable the validation of psychometric instruments in the specific population of parents of preterm infants. Also, the investigators can investigate the effect and predictive value of the course of parental depression, anxiety and stress scores on child's developmental outcome and on parent-infant bonding and attachment.

Thirdly, studies on epigenetic changes due to prenatal stress are still scarce in humans. In this study, the investigators will include a cohort of mothers experiencing profound prenatal stress due to preterm labor, which will complement the earlier work that has been carried out in a low-risk population. The investigators expect more profound changes in methylation state of the NR3C1 and other promotor regions in their cohort of mothers exposed to important prenatal stress. Secondly, the methylation of oxytocin receptor regions will be studied in relation to attachment and bonding.

An important overall goal of the project is to develop a Perinatal Stress Calculator that studies the value of the different neonatal, endocrinological, psychological and physiological stress-related parameters to predict differences in psychomotor, cognitive, behavioral, and emotional development. This longitudinal study design will enable the investigators to use the perinatal stress calculator to study the relation between the perinatal stress parameters and later developmental disabilities such as motor impairment, cognitive deficits, language delay but also social and behavioral problems such as attentional deficits and emotional self-regulation dysfunction.

DETAILED DESCRIPTION:
Project goals and their impact on societal challenges:

Objective 1: The first goal of the project is to identify objective stress markers that can be obtained easily and non-invasively in preterm infants during NICU hospitalization. This will include the development of novel techniques to measure stress related heart rate variability (HRV) and EEG maturation, as well as sleep stage markers. On a societal and economical level, reliable measures of the degree of distress in a hospitalized preterm infant will enable the evaluation of the direct effects of stress-reducing interventions such as NICU architecture changes and early intervention programs in cost benefit analyses. (Work package 1)

Objective 2: Second, the investigators aim to study the emotional and bonding processes in parents of preterm infants. Parental distress in terms of depressive symptoms, anxiety, perceived stress and parent-infant bonding will be measured at multiple time points. This will lead to the validation of psychometric instruments in the specific population of parents of preterm infants. Also, the investigators will investigate the effect and predictive value of the course of parental depression, anxiety and stress on children's developmental outcome and on parent-infant bonding and attachment. Knowledge about the short and long term risks of parental emotional distress are important to implement sufficient and tailored support to parents. (Work package 2)

Objective 3: Third, studies on epigenetic changes due to prenatal stress are still scarce in humans. Recently, preliminary evidence was found that prenatal stress affects the methylation state of the NR3C1promotor regions (Hompes et al., 2013). In this study, the investigators will include a cohort of mothers experiencing profound prenatal stress due to preterm labor, which will complement the earlier work that has been carried out in a low-risk population. The investigators expect more profound changes in methylation state of the NR3C1 and other promotor regions in this cohort. The methylation of oxytocin receptor genes will also be studied in relation to attachment and bonding. On a societal level, knowledge about the impact of adverse maternal psychological well-being during pregnancy on the epigenome is important, for example to justify prevention campaigns. (Work package 3)

Overall objective: An important overall goal of the project is to develop a Perinatal Stress Calculator that combines the values of the different neonatal, endocrinological, psychological and physiological stress-related parameters to predict differences in psychomotor, cognitive, behavioural, and emotional development (Work package 5). This prospective longitudinal study design will enable the investigators to use the perinatal stress calculator to study the relation between the perinatal stress parameters and later developmental disabilities such as motor impairment, cognitive deficits, and language delay but also social and behavioural problems such as attentional deficits and emotional self-regulation dysfunction (Work package 4). The investigators will not only be able to weigh perinatal infant characteristics in the model, but also parental characteristics such as distress, resilience and personality as well as bonding and attachment measures. On a societal and economic level, the results of the project will be important for health policy decision-making. Improved prediction of the developmental trajectory of preterm infants could lead to earlier and targeted interventions to decrease maladaptive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born before 34 weeks gestational age and/or with a birth weight lower than 1500g and their parents

Exclusion Criteria:

* Age < 18yr.
* Unable to speak and understand Dutch, French or English
* Unstable medical (somatic and/or psychiatric) disease in the parent(s)
* The presence of a major congenital malformation in the preterm infant

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The investigators will approach parents of preterm infants born before 34 weeks gestational age and/or with a birth weight lower than 1500g.
  Ideally, pregnant women admitted to the maternal intensive care (MIC) for preterm labor will be informed about the study together with their partner, and asked for consent. But in a number of preterm infants prenatal inclusion will not be possible (e.g. birth in another hospital, preterm premature rupture of the membranes,…) . Parents of infants in this subgroup, who are admitted to the Neonatal Intensive Care Unit (NICU) at the University Hospitals Leuven, will be informed and asked for consent within 3 days after birth.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2016-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Attachment behavior (will be assessed using questionnaires and both free and structured observations of the child-parent interaction) | 24 months

SECONDARY OUTCOMES:
Psychomotor development (will be assessed using Infant Scales of Development) | 24 months
Cognitive development (will be assessed using Infant Scales of Development) | 24 months
Cognitive development (executive functioning will be assessed by the Snack Delay Task) | 24 months
Language development (will be assessed using Infant Scales of Development) | 24 months
Language development (will be assessed using the NCDI-2A) | 24 months
Behavioral development (will be assessed using Infant Scales of Development ) | 24 months
Behavioral development (will be assessed by questioning both parents and external caregivers) | 24 months
Physical development (will be assessed by measuring children's height) | 24 months
Physical development (will be assessed by measuring children's weight) | 24 months
Physical development (will be assessed by measuring children's head circumference) | 24 months
Emotional development (will be assessed using the Bayley Scales of Infant Development III) | 24 months
Emotional development (will be assessed by questioning both parents and external caregivers) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Naulaers, MD, PhD, Principal Investigator — UZ / KU Leuven
Locations (1):
- UZLEUVEN, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aarnoudse-Moens CS, Weisglas-Kuperus N, van Goudoever JB, Oosterlaan J. Meta-analysis of neurobehavioral outcomes in very preterm and/or very low birth weight children. Pediatrics. 2009 Aug;124(2):717-28. doi: 10.1542/peds.2008-2816. Epub 2009 Jul 27. PMID 19651588
- [Background] Andre M, Lamblin MD, d'Allest AM, Curzi-Dascalova L, Moussalli-Salefranque F, S Nguyen The T, Vecchierini-Blineau MF, Wallois F, Walls-Esquivel E, Plouin P. Electroencephalography in premature and full-term infants. Developmental features and glossary. Neurophysiol Clin. 2010 May;40(2):59-124. doi: 10.1016/j.neucli.2010.02.002. Epub 2010 Mar 16. PMID 20510792
- [Background] Bosmans G, De Raedt R, Braet C. The invisible bonds: does the secure base script of attachment influence children's attention toward their mother? J Clin Child Adolesc Psychol. 2007 Oct-Dec;36(4):557-67. doi: 10.1080/15374410701662717. PMID 18088214
- [Background] Bosmans G, Braet C, Koster E, De Raedt R. Attachment security and attentional breadth toward the attachment figure in middle childhood. J Clin Child Adolesc Psychol. 2009 Nov;38(6):872-82. doi: 10.1080/15374410903258926. PMID 20183670
- [Background] Bowlby J, Attachment and Loss: Attachment V, Basic Books, 1969.
- [Background] Braeken MA, Kemp AH, Outhred T, Otte RA, Monsieur GJ, Jones A, Van den Bergh BR. Pregnant mothers with resolved anxiety disorders and their offspring have reduced heart rate variability: implications for the health of children. PLoS One. 2013 Dec 10;8(12):e83186. doi: 10.1371/journal.pone.0083186. eCollection 2013. PMID 24340091
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Carpenter LL, Carvalho JP, Tyrka AR, Wier LM, Mello AF, Mello MF, Anderson GM, Wilkinson CW, Price LH. Decreased adrenocorticotropic hormone and cortisol responses to stress in healthy adults reporting significant childhood maltreatment. Biol Psychiatry. 2007 Nov 15;62(10):1080-7. doi: 10.1016/j.biopsych.2007.05.002. Epub 2007 Jul 27. PMID 17662255
- [Background] Cassidy J. The nature of the child's ties. Handbook of attachment: Theory, research, and clinical implications 2:3-22, 1999.
- [Background] Cecchini M, Baroni E, Di Vito C, Piccolo F, Lai C. Newborn preference for a new face vs. a previously seen communicative or motionless face. Infant Behav Dev. 2011 Jun;34(3):424-33. doi: 10.1016/j.infbeh.2011.04.002. Epub 2011 May 8. PMID 21550665
- [Background] Chrousos GP. Stress and disorders of the stress system. Nat Rev Endocrinol. 2009 Jul;5(7):374-81. doi: 10.1038/nrendo.2009.106. Epub 2009 Jun 2. PMID 19488073
- [Background] Coolen MW, Statham AL, Gardiner-Garden M, Clark SJ. Genomic profiling of CpG methylation and allelic specificity using quantitative high-throughput mass spectrometry: critical evaluation and improvements. Nucleic Acids Res. 2007;35(18):e119. doi: 10.1093/nar/gkm662. Epub 2007 Sep 13. PMID 17855397
- [Background] Dykas MJ, Ehrlich KB, Cassidy J. Links between attachment and social information processing: examination of intergenerational processes. Adv Child Dev Behav. 2011;40:51-94. doi: 10.1016/b978-0-12-386491-8.00002-5. PMID 21887959
- [Background] Feldman R, Gordon I, Zagoory-Sharon O. Maternal and paternal plasma, salivary, and urinary oxytocin and parent-infant synchrony: considering stress and affiliation components of human bonding. Dev Sci. 2011 Jul;14(4):752-61. doi: 10.1111/j.1467-7687.2010.01021.x. Epub 2010 Dec 16. PMID 21676095
- [Background] Feldman R, Weller A, Zagoory-Sharon O, Levine A. Evidence for a neuroendocrinological foundation of human affiliation: plasma oxytocin levels across pregnancy and the postpartum period predict mother-infant bonding. Psychol Sci. 2007 Nov;18(11):965-70. doi: 10.1111/j.1467-9280.2007.02010.x. PMID 17958710
- [Background] Fisher DA. Thyroid system immaturities in very low birth weight premature infants. Semin Perinatol. 2008 Dec;32(6):387-97. doi: 10.1053/j.semperi.2008.09.003. PMID 19007675
- [Background] Gitau R, Fisk NM, Teixeira JM, Cameron A, Glover V. Fetal hypothalamic-pituitary-adrenal stress responses to invasive procedures are independent of maternal responses. J Clin Endocrinol Metab. 2001 Jan;86(1):104-9. doi: 10.1210/jcem.86.1.7090. PMID 11231985
- [Background] Glover V. Annual Research Review: Prenatal stress and the origins of psychopathology: an evolutionary perspective. J Child Psychol Psychiatry. 2011 Apr;52(4):356-67. doi: 10.1111/j.1469-7610.2011.02371.x. Epub 2011 Jan 19. PMID 21250994
- [Background] Glover V, O'Connor TG, O'Donnell K. Prenatal stress and the programming of the HPA axis. Neurosci Biobehav Rev. 2010 Sep;35(1):17-22. doi: 10.1016/j.neubiorev.2009.11.008. Epub 2009 Nov 13. PMID 19914282
- [Background] Heim C, Newport DJ, Bonsall R, Miller AH, Nemeroff CB. Altered pituitary-adrenal axis responses to provocative challenge tests in adult survivors of childhood abuse. Am J Psychiatry. 2001 Apr;158(4):575-81. doi: 10.1176/appi.ajp.158.4.575. PMID 11282691
- [Background] Heim C, Shugart M, Craighead WE, Nemeroff CB. Neurobiological and psychiatric consequences of child abuse and neglect. Dev Psychobiol. 2010 Nov;52(7):671-90. doi: 10.1002/dev.20494. PMID 20882586
- [Background] Hompes T, Izzi B, Gellens E, Morreels M, Fieuws S, Pexsters A, Schops G, Dom M, Van Bree R, Freson K, Verhaeghe J, Spitz B, Demyttenaere K, Glover V, Van den Bergh B, Allegaert K, Claes S. Investigating the influence of maternal cortisol and emotional state during pregnancy on the DNA methylation status of the glucocorticoid receptor gene (NR3C1) promoter region in cord blood. J Psychiatr Res. 2013 Jul;47(7):880-91. doi: 10.1016/j.jpsychires.2013.03.009. Epub 2013 Apr 6. PMID 23566423
- [Background] Izzi B, Decallonne B, Devriendt K, Bouillon R, Vanderschueren D, Levtchenko E, de Zegher F, Van den Bruel A, Lambrechts D, Van Geet C, Freson K. A new approach to imprinting mutation detection in GNAS by Sequenom EpiTYPER system. Clin Chim Acta. 2010 Dec 14;411(23-24):2033-9. doi: 10.1016/j.cca.2010.08.034. Epub 2010 Aug 31. PMID 20807523
- [Background] Kochanska G, Murray KT, Harlan ET. Effortful control in early childhood: continuity and change, antecedents, and implications for social development. Dev Psychol. 2000 Mar;36(2):220-32. PMID 10749079
- [Background] Lockwood CJ, Radunovic N, Nastic D, Petkovic S, Aigner S, Berkowitz GS. Corticotropin-releasing hormone and related pituitary-adrenal axis hormones in fetal and maternal blood during the second half of pregnancy. J Perinat Med. 1996;24(3):243-51. doi: 10.1515/jpme.1996.24.3.243. PMID 8827573
- [Background] McGowan PO, Sasaki A, D'Alessio AC, Dymov S, Labonte B, Szyf M, Turecki G, Meaney MJ. Epigenetic regulation of the glucocorticoid receptor in human brain associates with childhood abuse. Nat Neurosci. 2009 Mar;12(3):342-8. doi: 10.1038/nn.2270. PMID 19234457
- [Background] Meaney MJ, Szyf M, Seckl JR. Epigenetic mechanisms of perinatal programming of hypothalamic-pituitary-adrenal function and health. Trends Mol Med. 2007 Jul;13(7):269-77. doi: 10.1016/j.molmed.2007.05.003. Epub 2007 Jun 4. PMID 17544850
- [Background] Meyer-Lindenberg A, Tost H. Neural mechanisms of social risk for psychiatric disorders. Nat Neurosci. 2012 Apr 15;15(5):663-8. doi: 10.1038/nn.3083. PMID 22504349
- [Background] Mrdalj J, Pallesen S, Milde AM, Jellestad FK, Murison R, Ursin R, Bjorvatn B, Gronli J. Early and later life stress alter brain activity and sleep in rats. PLoS One. 2013 Jul 26;8(7):e69923. doi: 10.1371/journal.pone.0069923. Print 2013. PMID 23922857
- [Background] Mirescu C, Peters JD, Gould E. Early life experience alters response of adult neurogenesis to stress. Nat Neurosci. 2004 Aug;7(8):841-6. doi: 10.1038/nn1290. Epub 2004 Jul 25. PMID 15273691
- [Background] Oberlander TF, Weinberg J, Papsdorf M, Grunau R, Misri S, Devlin AM. Prenatal exposure to maternal depression, neonatal methylation of human glucocorticoid receptor gene (NR3C1) and infant cortisol stress responses. Epigenetics. 2008 Mar-Apr;3(2):97-106. doi: 10.4161/epi.3.2.6034. PMID 18536531
- [Background] Palmu K, Kirjavainen T, Stjerna S, Salokivi T, Vanhatalo S. Sleep wake cycling in early preterm infants: comparison of polysomnographic recordings with a novel EEG-based index. Clin Neurophysiol. 2013 Sep;124(9):1807-14. doi: 10.1016/j.clinph.2013.03.010. Epub 2013 Apr 30. PMID 23639376
- [Background] Patel J, Landers K, Li H, Mortimer RH, Richard K. Thyroid hormones and fetal neurological development. J Endocrinol. 2011 Apr;209(1):1-8. doi: 10.1530/JOE-10-0444. Epub 2011 Jan 6. PMID 21212091
- [Background] Pechtel P, Pizzagalli DA. Effects of early life stress on cognitive and affective function: an integrated review of human literature. Psychopharmacology (Berl). 2011 Mar;214(1):55-70. doi: 10.1007/s00213-010-2009-2. Epub 2010 Sep 24. PMID 20865251
- [Background] Reuss ML, Paneth N, Pinto-Martin JA, Lorenz JM, Susser M. The relation of transient hypothyroxinemia in preterm infants to neurologic development at two years of age. N Engl J Med. 1996 Mar 28;334(13):821-7. doi: 10.1056/NEJM199603283341303. PMID 8596548
- [Background] Reijneveld SA, de Kleine MJ, van Baar AL, Kollee LA, Verhaak CM, Verhulst FC, Verloove-Vanhorick SP. Behavioural and emotional problems in very preterm and very low birthweight infants at age 5 years. Arch Dis Child Fetal Neonatal Ed. 2006 Nov;91(6):F423-8. doi: 10.1136/adc.2006.093674. Epub 2006 Jul 28. PMID 16877476
- [Background] Sai FZ. The role of the mother's voice in developing mother's face preference: Evidence for intermodal perception at birth.
- [Background] Smith SL, Haley S, Slater H, Moyer-Mileur LJ. Heart rate variability during caregiving and sleep after massage therapy in preterm infants. Early Hum Dev. 2013 Aug;89(8):525-9. doi: 10.1016/j.earlhumdev.2013.01.004. Epub 2013 Jan 27. PMID 23361061
- [Background] Singer LT, Fulton S, Davillier M, Koshy D, Salvator A, Baley JE. Effects of infant risk status and maternal psychological distress on maternal-infant interactions during the first year of life. J Dev Behav Pediatr. 2003 Aug;24(4):233-41. doi: 10.1097/00004703-200308000-00003. PMID 12915795
- [Background] Spruyt A, Clarysse J, Vansteenwegen D, Baeyens F, Hermans D. Affect 4.0: a free software package for implementing psychological and psychophysiological experiments. Exp Psychol. 2010;57(1):36-45. doi: 10.1027/1618-3169/a000005. PMID 20178962
- [Background] Unternaehrer E, Luers P, Mill J, Dempster E, Meyer AH, Staehli S, Lieb R, Hellhammer DH, Meinlschmidt G. Dynamic changes in DNA methylation of stress-associated genes (OXTR, BDNF ) after acute psychosocial stress. Transl Psychiatry. 2012 Aug 14;2(8):e150. doi: 10.1038/tp.2012.77. PMID 22892716
- [Background] Van Beek Y, Hopkins B, Hoeksma JB. Development of communicative behaviors in preterm infants: The effects of birthweight status and gestational age. Infant Behavior and Development 17(2):107-117, 1994.
- [Background] Van Belle V, Neven P, Harvey V, Van Huffel S, Suykens JA, Boyd S. Risk group detection and survival function estimation for interval coded survival methods. Neurocomputing 112:200-210, 2013.
- [Background] Van Belle VM, Van Calster B, Timmerman D, Bourne T, Bottomley C, Valentin L, Neven P, Van Huffel S, Suykens JA, Boyd S. A mathematical model for interpretable clinical decision support with applications in gynecology. PLoS One. 2012;7(3):e34312. doi: 10.1371/journal.pone.0034312. Epub 2012 Mar 29. PMID 22479598
- [Background] Van den Bergh BR, Mennes M, Oosterlaan J, Stevens V, Stiers P, Marcoen A, Lagae L. High antenatal maternal anxiety is related to impulsivity during performance on cognitive tasks in 14- and 15-year-olds. Neurosci Biobehav Rev. 2005 Apr;29(2):259-69. doi: 10.1016/j.neubiorev.2004.10.010. Epub 2004 Dec 15. PMID 15811497
- [Background] Van den Bergh BR, Mulder EJ, Mennes M, Glover V. Antenatal maternal anxiety and stress and the neurobehavioural development of the fetus and child: links and possible mechanisms. A review. Neurosci Biobehav Rev. 2005 Apr;29(2):237-58. doi: 10.1016/j.neubiorev.2004.10.007. PMID 15811496
- [Background] van Londen WM, Juffer F, van Ijzendoorn MH. Attachment, cognitive, and motor development in adopted children: short-term outcomes after international adoption. J Pediatr Psychol. 2007 Nov-Dec;32(10):1249-58. doi: 10.1093/jpepsy/jsm062. Epub 2007 Aug 19. PMID 17709336
- [Background] van Putten MJ, Tavy DL. Continuous quantitative EEG monitoring in hemispheric stroke patients using the brain symmetry index. Stroke. 2004 Nov;35(11):2489-92. doi: 10.1161/01.STR.0000144649.49861.1d. Epub 2004 Oct 7. PMID 15472102
- [Background] Walton GE, Bower NJA, Bower TGR. Recognition of familiar faces by newborns. Infant Behavior and Development 15(2):265-269, 1992.
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608
- [Background] Bottomley C, Van Belle V, Mukri F, Kirk E, Van Huffel S, Timmerman D, Bourne T. The optimal timing of an ultrasound scan to assess the location and viability of an early pregnancy. Hum Reprod. 2009 Aug;24(8):1811-7. doi: 10.1093/humrep/dep084. Epub 2009 Apr 10. PMID 19363041
- [Background] Luts J., Molenberghs G., Verbeke G., Van Huffel S., Suykens J.A.K. A mixed effects least squares support vector machine model for classification of longitudinal data. Statistics & Data Analysis 56(3): 611-628, 2012.
- [Background] Vangeel EB, Izzi B, Hompes T, Vansteelandt K, Lambrechts D, Freson K, Claes S. DNA methylation in imprinted genes IGF2 and GNASXL is associated with prenatal maternal stress. Genes Brain Behav. 2015 Nov;14(8):573-82. doi: 10.1111/gbb.12249. Epub 2015 Sep 23. PMID 26333472
- [Background] Varrault A, Gueydan C, Delalbre A, Bellmann A, Houssami S, Aknin C, Severac D, Chotard L, Kahli M, Le Digarcher A, Pavlidis P, Journot L. Zac1 regulates an imprinted gene network critically involved in the control of embryonic growth. Dev Cell. 2006 Nov;11(5):711-22. doi: 10.1016/j.devcel.2006.09.003. PMID 17084362
- [Background] World Health Organization (2002). Iron and folate supplementation. Integrated management of pregnancy and childbirth (IMPAC). Standards for Maternal and Neonatal Care. http://www.who.int/reproductivehealth/publications/maternal_perinatal_health/iron_folate_supplementation.pdf The Department of Making Pregnancy Safer, World Health Organization.
- [Background] Feldman R, Gordon I, Zagoory-Sharon O. The cross-generation transmission of oxytocin in humans. Horm Behav. 2010 Sep;58(4):669-76. doi: 10.1016/j.yhbeh.2010.06.005. Epub 2010 Jun 15. PMID 20558167
- [Background] Feldman R, Gordon I, Schneiderman I, Weisman O, Zagoory-Sharon O. Natural variations in maternal and paternal care are associated with systematic changes in oxytocin following parent-infant contact. Psychoneuroendocrinology. 2010 Sep;35(8):1133-41. doi: 10.1016/j.psyneuen.2010.01.013. Epub 2010 Feb 12. PMID 20153585
- [Derived] Van den Brande A, Bollen B, Boets B, Naulaers G, Ortibus E. Executive Function Assessment in 2-Year-Olds Born Preterm. Neuropediatrics. 2024 Feb;55(1):16-22. doi: 10.1055/a-2023-9280. Epub 2023 Jan 31. PMID 36720262